CLINICAL TRIAL: NCT04234139
Title: Cohort/Ethics Study of Patients With Severe Alcoholic Hepatitis Undergoing Early Liver Transplantation
Status: Enrolling by invitation | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00154881; P50AA027054 (NIH)
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Liver Diseases, Alcoholic; Alcohol-Related Disorders; Transplant; Failure, Liver; Transplant; Complication, Rejection; Liver Diseases; Hepatitis, Alcoholic; Alcohol-Induced Disorders
Keywords: liver transplant; alcoholic liver disease
MeSH Terms: conditions — Liver Diseases, Alcoholic; Alcohol-Related Disorders; Rejection, Psychology; Liver Diseases; Hepatitis, Alcoholic; Alcohol-Induced Disorders | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective Cohort: Early Liver Transplantation (ELT) for patients who presented with Severe Alcoholic Hepatitis (SAH)
  Interventions: Procedure: liver transplant
- Prospective Cohort 1: Early Liver Transplantation (ELT) for patients who present with Severe Alcoholic Hepatitis (SAH)
  Interventions: Procedure: liver transplant
- Prospective Cohort 2: Orthotopic Liver Transplantation (OLT) in patient who present with Alcoholic Liver Disease (ALD)
  Interventions: Procedure: liver transplant

INTERVENTIONS:
Procedure: liver transplant — solid organ transplant

SUMMARY:
The purpose of this study is to develop a clinical understanding of early liver transplantation (ELT) for patients with severe alcoholic hepatitis (SAH) and identify the public's opinion regarding this practice.

DETAILED DESCRIPTION:
The research study is designed to improve the investigators' understanding of early liver transplantation for patients with severe alcoholic hepatitis. The goal of this research is twofold:

1. Establish a knowledge base necessary for appropriate liver transplant candidate selection by quantifying post-ELT mortality for SAH and compare to outcomes to liver transplantation for other indications
2. Develop an ethical framework for implementation of these transplants for SAH based on the opinions of healthcare providers and the general public.

ELIGIBILITY:
Inclusion Criteria for Severe Alcoholic Hepatitis patients:

* Patients with Severe Alcoholic Hepatitis (SAH) listed for liver transplantation at Johns Hopkins Hospital (JHH), have not been sober for at least 6 months at time of waitlisting, and are at least 18 years old.

Exclusion Criteria for Severe Alcoholic Hepatitis patients:

* Non-SAH patients listed for liver transplantation at JHH and patients who have been sober for at least 6 months at the time of waitlisting.

Inclusion Criteria for non-SAH comparison group:

* Patients 18 years or older undergoing liver transplantation at JHH for alcoholic liver disease and were sober for at least 6 months prior to transplantation.

Exclusion Criteria for non-SAH comparison group:

* Patients who do not meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe Alcoholic Hepatitis patients listed for liver transplatation at Johns Hopkins Hospital and patients undergoing liver transplantation at Johns Hopkins Hospital for Alcoholic Liver Disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who survived within 1 year post-transplant | 1 years
  Post-transplant survival within one year of the surgical procedure.

SECONDARY OUTCOMES:
Number of participants who self-report or have biochemically measured alcohol recidivism or relapse within 1 year post-transplant | 1 years
  Self-reported or biochemically measured alcohol recidivism or relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Cameron, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee BP, Chen PH, Haugen C, Hernaez R, Gurakar A, Philosophe B, Dagher N, Moore SA, Li Z, Cameron AM. Three-year Results of a Pilot Program in Early Liver Transplantation for Severe Alcoholic Hepatitis. Ann Surg. 2017 Jan;265(1):20-29. doi: 10.1097/SLA.0000000000001831. PMID 27280501
- [Background] Weeks SR, Sun Z, McCaul ME, Zhu H, Anders RA, Philosophe B, Ottmann SE, Garonzik Wang JM, Gurakar AO, Cameron AM. Liver Transplantation for Severe Alcoholic Hepatitis, Updated Lessons from the World's Largest Series. J Am Coll Surg. 2018 Apr;226(4):549-557. doi: 10.1016/j.jamcollsurg.2017.12.044. Epub 2018 Feb 2. PMID 29409981